CLINICAL TRIAL: NCT05030766
Title: A Pilot SMART Pre- and Post-testing of an Integrative Mindfulness-Based Smoking Cessation Intervention for HIV Patients
Brief Title: Testing Integrative Smoking Cessation for HIV Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Taghrid Asfar, Research Assistant Professor, University of Miami
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 20201296
Record Dates: First submitted 2021-08-26; First posted 2021-09-01 (Actual); Results first posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Smoking; Smoking Cessation; HIV Infections
Keywords: Mindfulness Training; Contingency Management
MeSH Terms: conditions — Smoking; Smoking Cessation; HIV Infections | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- MT plus NRT Group-Phase 1 (Experimental): Participants who receive the Mindfulness Training (MT) intervention for 4 weeks in addition to 6 weeks of Nicotine Replacement Therapy (NRT).These participants are responders (have quit smoking at the 1 month follow up) or non-responders (those who have not quit smoking at the 1 month follow up) and randomized to receive no additional intervention.
  Interventions: Drug: Nicotine Replacement Therapy; Behavioral: Mindfulness Training Smoking Cessation Intervention
- CM plus NRT Group-Phase1 (Experimental): Participants who receive the Contingency Management (CM) intervention for 4 weeks in addition to 6 weeks of NRT. These participants are responders (have quit smoking at the 1 month follow up) or non-responders (those who have not quit smoking at the 1 month follow up) and randomized to receive no additional intervention.
  Interventions: Drug: Nicotine Replacement Therapy; Behavioral: Contingency Management Smoking Cessation Intervention
- MT plus NRT with additional CM Group-Phase2 (Experimental): Participants who received the MT intervention for 4 weeks with 6 weeks of NRT and are non-responders (those who have not quit smoking at the 1 month follow up) and randomized to receive an additional CM intervention for another 4 weeks.
  Interventions: Drug: Nicotine Replacement Therapy; Behavioral: Mindfulness Training Smoking Cessation Intervention; Behavioral: Contingency Management Smoking Cessation Intervention
- CM plus NRT with additional MT Group-Phase2 (Experimental): Participants who received the CM intervention for 4 weeks with 6 weeks of NRT and are non-responders (those who have not quit smoking at the 1 month follow up) and randomized to receive an additional MT intervention for another 4 weeks.
  Interventions: Drug: Nicotine Replacement Therapy; Behavioral: Mindfulness Training Smoking Cessation Intervention; Behavioral: Contingency Management Smoking Cessation Intervention

INTERVENTIONS:
Drug: Nicotine Replacement Therapy — 6 weeks of Nicotine replacement patches
Behavioral: Mindfulness Training Smoking Cessation Intervention — Mindfulness Training Smoking Cessation Intervention administered online via Zoom. Each session lasts 60-90 minutes, twice weekly for 4 weeks for a total of 8 sessions.
  Arms: CM plus NRT with additional MT Group-Phase2; MT plus NRT Group-Phase 1; MT plus NRT with additional CM Group-Phase2
Behavioral: Contingency Management Smoking Cessation Intervention — Contingency Management Smoking Cessation Intervention includes one orientation session lasting about 60-90 minutes administered via Zoom. Participants will then be required to contact the research associate about their quitting progress three times a week for 4 weeks also by zoom.
  Arms: CM plus NRT Group-Phase1; CM plus NRT with additional MT Group-Phase2; MT plus NRT with additional CM Group-Phase2

SUMMARY:
The purpose of this study is to examine the feasibility, acceptability and effect of a combined smoking cessation intervention integrating contingency management (reward-based) strategies with Mindfulness training to identify the optimal dynamic strategy to promote smoking cessation among HIV patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HIV (based on self-report).
* Be 18 years and older
* Have smoked ≥ 5 cigarettes/day in the past year
* Be interested in making a quit attempt in the next 30 days
* Own a smartphone (apple/android), and plan to keep it active for the next 6 months
* Able to consent
* Have no plans to move in the next 6 months
* Are not pregnant or planning to be pregnant in the following 6 months
* Have any condition that, in the opinion of the investigator, would compromise the well-being of the patient or the study or prevent the patient from meeting or performing study requirements

Exclusion Criteria:

* Have contraindication to NRT (past month myocardial infarction, history of serious arrhythmias/or unstable angina pectoris, dermatological disorder)
* Are currently being treated for a psychiatric condition.
* Are currently being treated for smoking cessation, alcoholism, or illicit drug use
* Are adults unable to consent
* Are individuals who are not yet adults
* Are pregnant women
* Are prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taghrid A. Asfar, MD, MSPH, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase 2 participants are participants that did not quit smoking in their respective Phase 1 group, who were then assigned to the opposite group in Phase 2. Phase 1 MT participants who did not quit smoking go to Phase 2 CM, Phase 1 CM participants who did not quit smoking go to Phase 2 MT. Those participants who quit smoking do not get randomized again.
Groups:
- Mindfulness Training (MT) and NRT (Phase 1): Participants who receive the Mindfulness Training (MT) intervention for 4 weeks in addition to 6 weeks of Nicotine Replacement Therapy (NRT).These participants are responders (have quit smoking at the 1 month follow up) or non-responders (those who have not quit smoking at the 1 month follow up) and randomized to receive no additional intervention.
  Nicotine Replacement Therapy: 6 weeks of Nicotine replacement patches
  Mindfulness Training Smoking Cessation Intervention: Mindfulness Training Smoking Cessation Intervention administered online via Zoom. Each session lasts 60-90 minutes, twice weekly for 4 weeks for a total of 8 sessions.
- Contingency Management (CM) and NRT (Phase 1): Participants who receive the Contingency Management (CM) intervention for 4 weeks in addition to 6 weeks of NRT. These participants are responders (have quit smoking at the 1 month follow up) or non-responders (those who have not quit smoking at the 1 month follow up) and randomized to receive no additional intervention.
  Nicotine Replacement Therapy: 6 weeks of Nicotine replacement patches
  Contingency Management Smoking Cessation Intervention: Contingency Management Smoking Cessation Intervention includes one orientation session lasting about 60-90 minutes administered via Zoom. Participants will then be required to contact the research associate about their quitting progress three times a week for 4 weeks also by zoom.
- Mindfulness Training (MT) and NRT + Additional CM Group (Phase 2): Participants who received the MT intervention for 4 weeks with 6 weeks of NRT and are non-responders (those who have not quit smoking at the 1 month follow up) and randomized to receive an additional CM intervention for another 4 weeks.
  Nicotine Replacement Therapy: 6 weeks of Nicotine replacement patches
  Mindfulness Training Smoking Cessation Intervention: Mindfulness Training Smoking Cessation Intervention administered online via Zoom. Each session lasts 60-90 minutes, twice weekly for 4 weeks for a total of 8 sessions.
  Contingency Management Smoking Cessation Intervention: Contingency Management Smoking Cessation Intervention includes one orientation session lasting about 60-90 minutes administered via Zoom. Participants will then be required to contact the research associate about their quitting progress three times a week for 4 weeks also by zoom.
- Contingency Management (CM) and NRT + Additional MT Group (Phase 2): Participants who received the CM intervention for 4 weeks with 6 weeks of NRT and are non-responders (those who have not quit smoking at the 1 month follow up) and randomized to receive an additional MT intervention for another 4 weeks.
  Nicotine Replacement Therapy: 6 weeks of Nicotine replacement patches
  Mindfulness Training Smoking Cessation Intervention: Mindfulness Training Smoking Cessation Intervention administered online via Zoom. Each session lasts 60-90 minutes, twice weekly for 4 weeks for a total of 8 sessions.
  Contingency Management Smoking Cessation Intervention: Contingency Management Smoking Cessation Intervention includes one orientation session lasting about 60-90 minutes administered via Zoom. Participants will then be required to contact the research associate about their quitting progress three times a week for 4 weeks also by zoom.
Period: Phase 1 Participants
Arm/Group | Mindfulness Training (MT) and NRT (Phase 1) | Contingency Management (CM) and NRT (Phase 1) | Mindfulness Training (MT) and NRT + Additional CM Group (Phase 2) | Contingency Management (CM) and NRT + Additional MT Group (Phase 2)
Started | 49 | 46 | 0 | 0
Completed | 21 | 15 | 0 | 0
Not Completed | 28 | 31 | 0 | 0
Not completed — Lost to Follow-up | 12 | 22 | 0 | 0
Not completed — Did not attend sessions after being randomized | 16 | 9 | 0 | 0
Period: Phase 2 Participants
Arm/Group | Mindfulness Training (MT) and NRT (Phase 1) | Contingency Management (CM) and NRT (Phase 1) | Mindfulness Training (MT) and NRT + Additional CM Group (Phase 2) | Contingency Management (CM) and NRT + Additional MT Group (Phase 2)
Started | 0 | 0 | 12 | 10
Completed | 0 | 0 | 6 | 8
Not Completed | 0 | 0 | 6 | 2
Not completed — Lost to Follow-up | 0 | 0 | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Training (MT) and NRT (Phase 1) | Contingency Management (CM) and NRT (Phase 1) | Total
Number analyzed (Participants) | 49 | 46 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.54 (8.49) | 51.59 (11.63) | 53.07 (10.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 21 | 46
  Male | 24 | 25 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39 | 36 | 75
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 3 | 2 | 5
  Non-Hispanic Black | 35 | 33 | 68
  Hispanic | 10 | 10 | 20
  Asian/ Asian American / Pacific Islander | 0 | 0 | 0
  Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting 7-day Point-prevalence Abstinence
Description: Defined as self-report of not smoking in the past 7-days, not even a puff and confirmed by expired carbon monoxide (CO) level cutoff of < 8 ppm using a coVita iCO™ Smokerlyzer® and/or NicoTests saliva sample of ≤ 30 ng/mL.
Time Frame: 4 weeks (end of treatment), and 3 months
Population: Only those who participated in their treatment (completed at least one session).
Measure: Number; unit: participants
Arm/Group | Mindfulness Training (MT) and NRT (Phase 1) | Contingency Management (CM) and NRT (Phase 1) | Mindfulness Training (MT) and NRT + Additional CM Group (Phase 2) | Contingency Management (CM) and NRT + Additional MT Group (Phase 2)
Number analyzed (Participants) | 49 | 46 | 12 | 10
participants
  4 weeks (end of treatment): number analyzed (Participants) | 33 | 37 | 12 | 10
  4 weeks (end of treatment) | 8 | 12 | 3 | 2
  3 months: number analyzed (Participants) | 33 | 37 | 10 | 10
  3 months | 12 | 9 | 1 | 2

2. Secondary Outcome: Retention Rate
Description: Treatment specific retention rates reported as the percentage of participants who completed their final 3-month assessment divided by the total of participants enrolled.
Time Frame: 3 months
Population: All participants who enrolled and were randomized.
Measure: Number; unit: percentage of patients
Arm/Group | Mindfulness Training (MT) and NRT (Phase 1) | Contingency Management (CM) and NRT (Phase 1) | Mindfulness Training (MT) and NRT + Additional CM Group (Phase 2) | Contingency Management (CM) and NRT + Additional MT Group (Phase 2)
Number analyzed (Participants) | 49 | 46 | 12 | 10
percentage of patients | 42.83 | 32.61 | 50.00 | 80.00

3. Secondary Outcome: Treatment Specific Adherence Rates
Description: Defined as number of phone-call check-ins attended by each participant (4 for mindfulness training, 12 for contingency management).
Time Frame: 3 months
Population: Includes all participants who were randomized to a treatment arm. Note that Phase 1 and Phase 2 participants are not mutually exclusive (Phase 2 participants come from Phase 1). Mindfulness Training participants did one call per week of treatment, 4 calls in total. Contingency management did 3 calls per week of treatment for a total of 12 calls.
Measure: Number; unit: participants
Arm/Group | Mindfulness Training (MT) and NRT (Phase 1) | Contingency Management (CM) and NRT (Phase 1) | Mindfulness Training (MT) and NRT + Additional CM Group (Phase 2) | Contingency Management (CM) and NRT + Additional MT Group (Phase 2)
Number analyzed (Participants) | 49 | 46 | 12 | 10
participants
  0 check-ins | 18 | 15 | 1 | 0
  Less than half the check-ins | 4 | 21 | 9 | 1
  Half of the check-ins | 2 | 5 | 0 | 1
  More than half the check-ins but did not complete all | 9 | 5 | 2 | 4
  Completed all check-ins | 16 | 0 | 0 | 4

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Mindfulness Training (MT) and NRT (Phase 1) | Contingency Management (CM) and NRT (Phase 1) | Mindfulness Training (MT) and NRT + Additional CM Group (Phase 2) | Contingency Management (CM) and NRT + Additional MT Group (Phase 2)
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/46 | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/46 | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 0/49 | 0/46 | 0/12 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-09): https://cdn.clinicaltrials.gov/large-docs/66/NCT05030766/Prot_SAP_000.pdf